CLINICAL TRIAL: NCT02323048
Title: Acquisition of Responses to a Methamphetamine-associated Cue in Healthy Humans: Self-report, Behavioral, and Psychophysiological Measures.
Brief Title: Acquisition of Responses to a Methamphetamine-associated Cue in Healthy Humans
Acronym: CAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 12-2047
Record Dates: First submitted 2014-10-30; First posted 2014-12-23 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Methamphetamine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Paired, high reward (Experimental): All participants will be administered methamphetamine (20mg) and placebo. All subjects received methamphetamine (20 mg) on two conditioning sessions and placebo on the other two sessions, administered under double-blind conditions.
  Interventions: Drug: methamphetamine; Drug: placebo
- Paired, low reward (Experimental): All participants will be administered methamphetamine (20mg) and placebo. All subjects received methamphetamine (20 mg) on two conditioning sessions and placebo on the other two sessions, administered under double-blind conditions.
  Interventions: Drug: methamphetamine; Drug: placebo
- Paired no reward (Experimental): All participants will be administered methamphetamine (20mg) and placebo. All subjects received methamphetamine (20 mg) on two conditioning sessions and placebo on the other two sessions, administered under double-blind conditions.
  Interventions: Drug: methamphetamine; Drug: placebo
- Unpaired, high reward (Experimental): All participants will be administered methamphetamine (20mg) and placebo. All subjects received methamphetamine (20 mg) on two conditioning sessions and placebo on the other two sessions, administered under double-blind conditions.
  Interventions: Drug: methamphetamine; Drug: placebo
- Unpaired, low reward (Experimental): All participants will be administered methamphetamine (20mg) and placebo. All subjects received methamphetamine (20 mg) on two conditioning sessions and placebo on the other two sessions, administered under double-blind conditions.
  Interventions: Drug: methamphetamine; Drug: placebo

INTERVENTIONS:
Drug: methamphetamine — : Twenty milligrams of MA (Desoxyn; Lundbeck Inc) tablets will be crushed and placed in 10 ml of Ora-Sweet syrup. Placebo drinks will consist of 10 ml of Ora-Sweet alone.
  Other Names: desoxyn
Drug: placebo — Placebo (sugar pill)
  Other Names: dextrose

SUMMARY:
The aim of the study is to extend our investigations of drug-associated conditioning with healthy volunteers. The investigators have recently completed a pilot study demonstrating that subjects show an increase in self-reported preference for a visual stimulus paired with stimulant drug administration. Furthermore, our pilot data suggest that methamphetamine acts synergistically with rewards in the environment, such that this conditioning effect is facilitated by experiencing the drug in the presence of rewarding, or positive events, such as earning money. The investigators now aim to extend these findings by assessing not only self-reported preference, but also attentional and psychophysiological (electromyogram; EMG) responses to the drug-associated stimuli.

DETAILED DESCRIPTION:
The study will consist of an orientation session following by 6 experimental study sessions. The first experimental session will consist of a "Pre-test", where baseline data regarding attentional, psychophysiological, and self-reported responses tovarious stimuli will be collected. The following 4 sessions will consist of a drug (sedative or stimulant) or placebo. During these sessions, subjects will play simple computer games, as well as complete questionnaires regarding mood and potential subjective drug effects. The subjects will then complete a "Test" session, where attentional, psychophysiological, and self-reported responses to the stimuli will be assessed, as in the first experimental session.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 19-26kg/m, high school education,
* fluency in English,
* resting blood pressure less than140/90mmHg and consumption of less than 4 standard alcohol or caffeinated drinks per day.

Exclusion Criteria:

* current substance abuse or lifetime substance dependence,
* regular medication,
* history of cardiovascular illness,
* current major Axis I DSM-IV disorder (APA, 2004),
* mood disorder or psychotic symptoms within the past year.
* Shift workers and pregnant or nursing mothers will also be excluded.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leah Mayo, Study Director — Graduate Student

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers aged 18-35 were recruited through posters, online and newspaper advertisement, and word-of mouth referrals throughout the community.
Groups:
- Paired, High Reward: All participants will be administered methamphetamine (20mg) and placebo. methamphetamine: : Twenty milligrams of MA (Desoxyn; Lundbeck Inc) tablets will be crushed and placed in 10 ml of Ora-Sweet syrup. Placebo drinks will consist of 10 ml of Ora-Sweet alone.
  placebo: Placebo (sugar pill)
  placebo: Placebo (sugar pill)
- Paired, Low Reward; Paired, no Reward; Unpaired, High Reward; Unpaired, Low Reward: All participants will be administered methamphetamine (20mg) and placebo. methamphetamine: : Twenty milligrams of MA (Desoxyn; Lundbeck Inc) tablets will be crushed and placed in 10 ml of Ora-Sweet syrup. Placebo drinks will consist of 10 ml of Ora-Sweet alone.
  placebo: Placebo (sugar pill)
Period: Overall Study
Arm/Group | Paired, High Reward | Paired, Low Reward | Paired, no Reward | Unpaired, High Reward | Unpaired, Low Reward
Started | 25 | 26 | 23 | 7 | 9
Completed | 24 | 24 | 23 | 7 | 9
Not Completed | 1 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers aged 18-35 with BMI between 19 and 26kg/m2, at least high school completed educated., resting bp less than 140/90, current alcohol consumption less than 4 drinks per day, less than 4 caffenated beverages per day. No major DSM IV disorder, no current psychoactive medication, no pregnancy
Groups:
- Paired, High Reward; Paired, Low Reward; Paired, no Reward; Unpaired, High Reward; Unpaired, Low Reward: All participants will be administered methamphetamine (20mg) and placebo.
  methamphetamine: : Twenty milligrams of MA (Desoxyn; Lundbeck Inc) tablets will be crushed and placed in 10 ml of Ora-Sweet syrup. Placebo drinks will consist of 10 ml of Ora-Sweet alone.
  placebo: Placebo (sugar pill)
- Total: Total of all reporting groups
Arm/Group | Paired, High Reward | Paired, Low Reward | Paired, no Reward | Unpaired, High Reward | Unpaired, Low Reward | Total
Number analyzed (Participants) | 24 | 24 | 23 | 7 | 9 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 23 | 7 | 9 | 87
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (5.0) | 23.9 (3.3) | 22.8 (2.3) | 23.3 (3.0) | 24.2 (3.7) | 23.8 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 13 | 5 | 4 | 49
  Male | 12 | 9 | 10 | 2 | 5 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 23 | 7 | 9 | 87

OUTCOME MEASURES:

1. Primary Outcome: Subjective Effects as Assessed by Score on "Feel Drug", "Feel High", "Like Drug", and "Want More" Subscales of the Drug Effects Questionnaire
Description: The Drug Effects Questionnaire (DEQ) is a visual analog scale questionnaire that assesses the extent to which subjects experience four subjective states: "Feel Drug", "Feel High", "Like Drug", and "Want More". The "Feel Drug", "Feel High", "Like Drug", and "Want More" subscales are reported. All subscales are scored on a visual analogue scale (scroll bar on computer screen) ranging from 0-100. 100 represents the highest score for that subjective state, and the higher the score, the worse the outcome.
Time Frame: End of study (time 0 and approximately 4 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Paired, High Reward (Methamphetamine Sessions); Paired, Low Reward (Methamphetamine Sessions); Paired no Reward (Methamphetamine Sessions); Unpaired, High Reward (Methamphetamine Sessions); Unpaired, Low Reward (Methamphetamine Sessions): All subjects received methamphetamine (20 mg) on two conditioning sessions
Arm/Group | Paired, High Reward (Methamphetamine Sessions) | Paired, Low Reward (Methamphetamine Sessions) | Paired no Reward (Methamphetamine Sessions) | Unpaired, High Reward (Methamphetamine Sessions) | Unpaired, Low Reward (Methamphetamine Sessions)
Number analyzed (Participants) | 24 | 24 | 23 | 7 | 9
units on a scale
  Feel Drug | 50.39 (3.29) | 45.25 (3.0) | 41.22 (2.5) | 48.55 (2.6) | 42.22 (2.5)
  Like Drug | 68.85 (3.32) | 64.25 (3.10) | 60.55 (3.0) | 61.55 (3.5) | 60.2 (3.4)
  Feel High | 42.04 (3.79) | 41.04 (3.55) | 38.88 (3.45) | 39.55 (3.45) | 38.0 (3.42)
  Want More | 65.11 (3.98) | 62.44 (3.55) | 61.55 (3.44) | 60.55 (3.42) | 59.5 (3.10)

ADVERSE EVENTS:
Arm/Group | Paired, No Reward | Paired, Low Reward | Paired, High Reward | Unpaired, Low Reward | Unpaired, High Reward
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/24 | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes